CLINICAL TRIAL: NCT04247815
Title: A Phase 2a, Randomized, Investigator and Patient-blind, Sponsor-unblinded, Parallel Group, Placebo-controlled Study of ATI-450 Plus Methotrexate (MTX) vs MTX Alone in Patients With Moderate to Severe Active Rheumatoid Arthritis
Brief Title: Study of ATI-450 Plus Methotrexate (MTX) vs MTX Alone in Patients With Moderate to Severe RA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATI-450-RA-201
Record Dates: First submitted 2020-01-16; First posted 2020-01-30 (Actual); Results first posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Arthritis; Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — Methotrexate

STUDY DESIGN:
Intervention Model Description: Randomized, investigator and patient-blind, sponsor-unblinded, parallel group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The blinded placebo drug is packaged to match the active study drug and will be stored under the same conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ATI-450 plus Methotrexate (Experimental): ATI-450 50mg oral tablet BID with a stable weekly dose of Methotrexate
  Interventions: Drug: ATI-450; Drug: Methotrexate
- Placebo plus Methotrexate (Placebo Comparator): Placebo oral tablet BID with a stable weekly dose of Methotrexate
  Interventions: Drug: Placebo oral tablet; Drug: Methotrexate

INTERVENTIONS:
Drug: ATI-450 — Oral, small molecule MK2 inhibitor
  Other Names: CDD-450
  Arms: ATI-450 plus Methotrexate
Drug: Placebo oral tablet — Placebo tablet manufactured to match ATI-450 in appearance
  Arms: Placebo plus Methotrexate
Drug: Methotrexate — 7.5 mg to 25 mg weekly

SUMMARY:
This is a Phase 2 study to investigate the safety, tolerability, PK, and PD of ATI-450 plus methotrexate versus methotrexate alone in patients with moderate to severe RA.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, investigator and patient-blind, sponsor-unblinded, parallel group, placebo-controlled study to investigate the safety, tolerability, PK, and PD of ATI-450 plus methotrexate versus methotrexate alone in patients with moderate to severe RA with inadequate response to methotrexate. All subjects will be required to complete a safety follow up visit 30 days post last study medication administration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adult-onset RA as defined by the 2010 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) classification criteria.
* DAS28-CRP ≥3.2 defined as moderate to high disease activity.
* Have moderately to severely active RA defined by at least 4/28 tender and 4/28 swollen joints.
* hsCRP ≥5 mg/L at screening.
* Patients must have definitive intra-articular synovitis or osteitis defined as a score of 1 or greater on a Hand-Wrist MRI as assessed by central imaging reader (using RAMRIS).
* On a stable MTX dose and a stable dose of folic or folinic acid prior to the screening visit.

Exclusion Criteria:

* Patient has a current acute or chronic immunoinflammatory disease other than RA which may impact the course or assessment of RA.
* Patient has an uncontrolled non-immunoinflammatory disease that may place the patient at increased risk during the study or impact the interpretation of results.
* History or evidence of active or latent tuberculosis.
* Active infection requiring treatment with antibiotics.
* Blood pressure levels (in supine position after at least 5 minutes rest): <90 mmHg or >140 mmHg for systolic blood pressure or <40 mmHg or >90 mmHg for diastolic blood pressure.
* Are currently receiving corticosteroids at doses greater than 10 mg per day of prednisone (or equivalent) or have been receiving an unstable dosing regimen of corticosteroids within 2 weeks of the screening visit.
* Have started treatment with non-steroidal anti-inflammatory drugs (NSAIDs) or have been receiving an unstable dosing regimen of NSAIDs within 2 weeks of the screening visit.
* Patients with history of stroke.
* Any joint procedure in the past 90 days prior to screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Gordon, Study Director — Aclaris Therapeutics
Locations (5):
- United States (5):
  - Aclaris Investigational Site, Anniston, Alabama
  - Aclaris Investigational Site, Tampa, Florida
  - Aclaris Investigational Site, Atlanta, Georgia
  - Aclaris Investigational Site, Duncansville, Pennsylvania
  - Aclaris Investigational Site, Mesquite, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ATI-450 Plus Methotrexate | Placebo Plus Methotrexate
Started | 16 | 3
Completed | 14 | 2
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ATI-450 Plus Methotrexate | Placebo Plus Methotrexate | Total
Number analyzed (Participants) | 16 | 3 | 19
Age, Customized [Mean (Standard Deviation); unit: years] | 55.9 (9.93) | 55.3 (6.81) | 55.8 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 3 | 14
  Male | 5 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 12 | 3 | 15
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 3 | 19
Weight (kg) [Mean (Standard Deviation); unit: kg] | 92.74 (25.504) | 98.93 (14.616) | 93.72 (23.899)
Height (cm) [Mean (Standard Deviation); unit: cm] | 166.94 (12.648) | 164.43 (3.092) | 166.54 (11.630)
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 33.37 (8.829) | 36.53 (4.737) | 33.87 (8.298)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure is the Determination of the Safety and Tolerability of ATI-450 Plus Methotrexate in Patients With Moderate to Severe Rheumatoid Arthritis: Adverse Events (AEs)
Description: Safety and tolerability reported as Adverse Events (AEs). AEs will be coded with the Medical Dictionary for Regulatory Activities (MedDRA) version 23.0. AEs will be presented by system organ class and preferred term in frequency tables.
Time Frame: Baseline through Day 114
Population: The Safety population consisted of patients who receive at least 1 dose of study drug. This set was used for the safety data summaries and baseline characteristic summaries. This set was analyzed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-450 Plus Methotrexate | Placebo Plus Methotrexate
Number analyzed (Participants) | 16 | 3
Participants | 8 | 2

2. Secondary Outcome: Percent Change in (hsCRP) Levels Over Time
Description: Median percent change from baseline in high sensitivity C-reactive protein (hsCRP) levels over time
Time Frame: Baseline through Day 114
Population: The Per-Protocol (PP) population consisted of all patients who completed their Day 84 visit and had valid hsCRP values for at least 6 of the 7 scheduled collection times. This set was analyzed as treated.
Measure: Median (Full Range); unit: Percent Change from Baseline hsCRP
Arm/Group | ATI-450 Plus Methotrexate | Placebo Plus Methotrexate
Number analyzed (Participants) | 15 | 2
Percent Change from Baseline hsCRP
  Week 1 | -75.00 [-97.3 to 11] | -16.50 [-34.9 to 1.9]
  Week 2: number analyzed (Participants) | 14 | 2
  Week 2 | -72.40 [-96.3 to 129.4] | 15.50 [-66.7 to 97.7]
  Week 4 | -51.10 [-96.6 to 285.3] | -50.20 [-81.2 to -19.2]
  Week 6 | -57.60 [-96.6 to 306.2] | 3.00 [-29.2 to 35.2]
  Week 8 | -74.20 [-92.9 to 63.3] | 78.50 [9.6 to 147.4]
  Week 12 | -42.60 [-97 to 263.7] | 7.30 [-5.6 to 20.2]
  Follow-up: number analyzed (Participants) | 14 | 2
  Follow-up | -15.60 [-83.1 to 143.2] | -40.65 [-66.7 to -14.6]

3. Secondary Outcome: Change From Baseline in Disease Activity Score
Description: The Disease Activity Score using 28 joint count C-reactive protein DAS28 (CRP) consists of a composite score of the following variables: tender joint count, swollen joint count, CRP, and Patient's Global Assessment of Disease Activity score.
  The following equation will be used to calculate the DAS28 (CRP):
  DAS28 (CRP) = 0.56 √TJC28 + 0.28√SJC28 + 0.36ln(CRP +1) + 0.014×(Patient's Global Assessment of Disease Activity) + 0.96, where:
  * TJC28 = number of joints tender out of 28
  * SJC28 = number of joints swollen out of 28
  * CRP = C-reactive protein
  * Patient's Global Assessment of Disease Activity on a 100 mm visual analog scale (VAS) recorded by the patient
  Interpretation of the DAS28 (CRP) disease activity measure is on a scale of 0 to 9.4, where: <2.6 is considered remission, ≥2.6 to <3.2 is considered low/minimal, ≥3.2 to ≤5.1 is considered moderate, and >5.1 is considered high/severe.
Time Frame: Baseline through Day 114
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATI-450 Plus Methotrexate | Placebo Plus Methotrexate
Number analyzed (Participants) | 15 | 2
score on a scale
  Baseline | 5.72 (0.970) | 6.00 (0.990)
  Week 1 | 4.33 (1.611) | 6.15 (0.495)
  Week 2: number analyzed (Participants) | 14 | 2
  Week 2 | 4.26 (1.570) | 5.25 (0.354)
  Week 4 | 4.11 (1.351) | 5.75 (1.061)
  Week 6 | 4.25 (1.436) | 6.15 (0.495)
  Week 8 | 3.84 (1.383) | 6.20 (0.424)
  Week 12 | 3.70 (1.574) | 6.35 (0.212)
  Follow-up: number analyzed (Participants) | 14 | 2
  Follow-up | 4.21 (1.705) | 4.95 (0.495)

4. Secondary Outcome: Number and Percent of Patients Achieving DAS28-CRP <2.6 Over Time
Description: Number and Percent of Patients Achieving DAS28-CRP <2.6 over time
Time Frame: Baseline through Day 114
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-450 Plus Methotrexate | Placebo Plus Methotrexate
Number analyzed (Participants) | 15 | 2
Participants
  Baseline | 0 | 0
  Week 1 | 2 | 0
  Week 2: number analyzed (Participants) | 14 | 2
  Week 2 | 3 | 0
  Week 4 | 2 | 0
  Week 6 | 1 | 0
  Week 8 | 2 | 0
  Week 12 | 3 | 0
  Follow-up: number analyzed (Participants) | 14 | 2
  Follow-up | 4 | 0

5. Secondary Outcome: Change From Baseline in RAMRIS Hand-Wrist Assessments (Osteitis Average)
Description: Rheumatoid Arthritis Magnetic Resonance Imaging Score (RAMRIS) uses integer scales to measure the severity of disease at each bone or joint of interest in the hand and wrist, with separate scores given for osteitis and synovitis.
  Osteitis was scored at 25 bone locations: distal radius and ulna, 8 carpal bones (trapezium, trapezoid, capitate, hamate, pisiform, scaphoid, lunate, and triquetrum, as well as the 5 metacarpal bases), 5 metacarpal heads, and 5 proximal phalangeal bases.
  Score Definition
  0 No osteitis
  1. 1-33% involvement of original articular bone
  2. 34-67% involvement of original articular bone
  3. 68-100% involvement of original articular bone
  Synovitis was scored at the following 8 joint locations: distal radioulnar joint, radiocarpal joint, intercarpal / carpometacarpal joints 2-5, and 5 metacarpophalangeal (MCP) joints.
  Score Definition
  0 No synovitis
  1. 1-33% volume enhancement
  2. 34-67% volume enhancement
  3. 68-100% volume enhancement
Time Frame: Baseline through Day 84
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Change in Osteitis average
Arm/Group | ATI-450 Plus Methotrexate | Placebo Plus Methotrexate
Number analyzed (Participants) | 15 | 2
Change in Osteitis average | 0.97 (1.943) | 0.88 (1.237)

6. Secondary Outcome: Change From Baseline in RAMRIS Hand-Wrist Assessments (Synovitis Average)
Description: as for outcome 5
Time Frame: Baseline through Day 84
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Change in Synovitis average
Arm/Group | ATI-450 Plus Methotrexate | Placebo Plus Methotrexate
Number analyzed (Participants) | 15 | 2
Change in Synovitis average | 0.08 (1.894) | 1.50 (2.121)

7. Secondary Outcome: Number and Percent of Patients Achieving ACR 20
Description: American College of Rheumatology (ACR) 20 will be calculated at each treatment visit and the number and percent of subjects with a 20% improvement will be tabulated at each scheduled visit.
Time Frame: Baseline through Day 114
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-450 Plus Methotrexate | Placebo Plus Methotrexate
Number analyzed (Participants) | 15 | 2
Participants
  Week 4 | 8 | 0
  Week 8 | 8 | 0
  Week 12 | 9 | 0
  Follow-up | 6 | 1

8. Secondary Outcome: Number and Percent of Patients Achieving ACR 50
Description: American College of Rheumatology (ACR) 50 will be calculated at each treatment visit and the number and percent of subjects with a 50% improvement will be tabulated at each scheduled visit.
Time Frame: Baseline through Day 114
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-450 Plus Methotrexate | Placebo Plus Methotrexate
Number analyzed (Participants) | 15 | 2
Participants
  Week 4 | 2 | 0
  Week 8 | 4 | 0
  Week 12 | 5 | 0
  Follow-up | 3 | 0

9. Secondary Outcome: Number and Percent of Patients Achieving ACR 70
Description: American College of Rheumatology (ACR) 70 will be calculated at each treatment visit and the number and percent of subjects with a 70% improvement will be tabulated at each scheduled visit.
Time Frame: Baseline through Day 114
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-450 Plus Methotrexate | Placebo Plus Methotrexate
Number analyzed (Participants) | 15 | 2
Participants
  Week 4 | 0 | 0
  Week 8 | 3 | 0
  Week 12 | 3 | 0
  Follow-up | 0 | 0

10. Secondary Outcome: Assessment of ATI-450 Concentration (ng/mL)
Time Frame: Day 1 through Day Day 84
Population: The PK population consisted of all patients who received at least 1 dose of study drug and provided at least 1 plasma concentration value. This set was analyzed as treated.
Measure: Mean (Standard Deviation); unit: ATI-450 concentration (ng/mL)
Arm/Group | ATI-450 Plus Methotrexate
Number analyzed (Participants) | 16
ATI-450 concentration (ng/mL)
  Day 1 (2 Hours Postdose): number analyzed (Participants) | 15
  Day 1 (2 Hours Postdose) | 225.87 (78.603)
  Day 7 (Predose) | 163.97 (85.538)
  Day 14 (Predose): number analyzed (Participants) | 15
  Day 14 (Predose) | 131.51 (55.175)
  Day 28 (Predose) | 135.67 (84.454)
  Day 42 (Predose): number analyzed (Participants) | 15
  Day 42 (Predose) | 170.84 (99.863)
  Day 56 (Predose): number analyzed (Participants) | 15
  Day 56 (Predose) | 153.45 (89.092)
  Day 84 (Predose) | 124.71 (69.437)
  Day 84 (2 Hours Postdose): number analyzed (Participants) | 14
  Day 84 (2 Hours Postdose) | 293.00 (98.643)

ADVERSE EVENTS:
Time Frame: Baseline to Day 114
Arm/Group | ATI-450 Plus Methotrexate | Placebo Plus Methotrexate
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/3
Other Adverse Events (participants affected / at risk) | 8/16 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATI-450 Plus Methotrexate (N=16) | Placebo Plus Methotrexate (N=3)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) — SAE occurred during the follow-up period.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATI-450 Plus Methotrexate (N=16) | Placebo Plus Methotrexate (N=3)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary tract infection (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0)
Low density lipoprotein increased (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/15/NCT04247815/Prot_SAP_002.pdf